CLINICAL TRIAL: NCT02857777
Title: An Open-Label, Single-Ascending Dose Study to Assess the Pharmacokinetics, Safety, and Tolerability of Intranasally Administered Esketamine in Elderly (>=65 Years of Age) Japanese, and Healthy Younger Adult Japanese Subjects (20 to 55 Years of Age, Inclusive)
Brief Title: Pharmacokinetic, Safety, and Tolerability Study of Intranasally Administered Esketamine in Elderly Japanese, and Healthy Younger Adult Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108213; 54135419TRD1018 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-08-03; First posted 2016-08-05 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — Esketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1: Japanese elderly subjects (Esketamine) (Experimental): Subjects will receive Treatment A (28 milligram [mg] of esketamine, administered as 1*14 mg spray of esketamine in each nostril at Time 0) in Period 1, Treatment B (56 mg of esketamine, administered as 1*14 mg spray of esketamine in each nostril at Time 0 and 5 minutes) in Period 2 and then Treatment C (84 mg of esketamine, administered as 1*14 mg spray of esketamine in each nostril at Time 0, 5, and 10 minutes) in Period 3. A washout period of 5 to 14 days will separate each intranasal esketamine treatment regimen.
  Interventions: Drug: Esketamine
- Cohort 2: Japanese healthy subjects (Esketamine) (Active Comparator): Subjects will receive Treatment A in Period 1, Treatment B in Period 2 and then Treatment C in Period 3. A washout period of 5 to 14 days will separate each intranasal esketamine treatment regimen.
  Interventions: Drug: Esketamine

INTERVENTIONS:
Drug: Esketamine — Subjects will self-administer intranasal esketamine as per the treatment regimen.

SUMMARY:
The purpose of this study is to compare the pharmacokinetics, safety, and tolerability of intranasally administered esketamine in elderly Japanese subjects and healthy younger adult Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* A) Cohort 1: Be a Japanese man or woman greater than or equal to (>=) 65 years of age with at least 4 subjects >= 70 years of age, who was born in Japan, who has resided outside of Japan for >= 10 years, with parents and maternal and paternal grandparents who are of Japanese ethnicity. Subjects must be either healthy or present with stable, well-controlled, chronic conditions which frequently occur in the elderly, such as: Hyperlipidemia,Controlled hypertension, Impaired fasting glucose, impaired glucose tolerance, or type 2 diabetes mellitus controlled with diet, and/or metformin monotherapy, dipeptidyl peptidase-4 (DPP-4) inhibitor monotherapy or a combination of metformin and DPP-4 inhibitor, who have glycated hemoglobin (HbA1c) levels <8 percent (%), Degenerative joint disorders and osteoporosis; B) Cohort 2: Be a healthy Japanese man or woman 20 to 55 years of age, inclusive, who was born in Japan, who has resided outside of Japan for >= 10 years, and has parents and maternal and paternal grandparents who are of Japanese ethnicity. Each subject will be matched to an elderly subject in Cohort 1 by gender and body weight (+/- 20%) using data collected during Screening
* Signed an informed consent document indicating they understand the purpose of and procedures required for the study and are willing to participate in the study
* Willing to adhere to the prohibitions and restrictions specified in this protocol
* Cohort 2: If a woman, must have a negative serum beta-human chorionic gonadotropin (hCG) pregnancy test at screening and a negative urine pregnancy test on Day -1 of the treatment period. Women using contraceptives must agree to use an additional birth control method during the study and for 1 month after receiving the last dose of study drug
* If a woman, must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction

Exclusion Criteria:

* Current significant psychiatric disorder including but not limited to psychotic, bipolar, major depressive, or anxiety disorder
* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the subject or that could interfere with the interpretation of the study results. Elderly subjects in Cohort 1 with stable, well-controlled, chronic conditions which frequently occur in the elderly as outlined in Inclusion Criteria 1 will be permitted to participate in the study
* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening or Day -1 of Period 1 as deemed appropriate by the investigator
* Clinically significant abnormal physical examination, vital signs, or 12 lead electrocardiogram (ECG) at screening or before the first study drug administration as deemed appropriate by the investigator
* History of moderate or severe use disorder according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-5) criteria within 1 year before screening or positive test result(s) for alcohol and/or drugs of abuse (such as barbiturates, opiates, cocaine, cannabinoids, amphetamines, and benzodiazepines) at screening and Day -1 of the treatment period

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-08-09 (Actual); Primary Completion 2017-01-27 (Actual); Study Completion 2017-01-27 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | up to Day 2
  The Cmax is the maximum plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to 12 hours (AUC [0-12]) | up to Day 2
  The AUC (0-12) is the area under the plasma concentration-time curve from time zero to 12 hours, calculated as the sum of AUC(last) and C(last)/lambda(z), wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time; and C(last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-last]) | up to Day 2
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time, calculated as the sum of AUC(last) and C(last)/lambda(z), wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time; and C(last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | up to Day 2
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z), wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time; and C(last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Terminal Half-Life(t[1/2]) | up to Day 2
  Terminal half-life (t[(1/2]) is defined as 0.693/Lambda(z).
Lambda(z) | up to Day 2
  Lambda(z) is the first-order rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Number of subjects with Adverse Events (AEs) as a measure of safety and tolerability | Screening up to Follow-up (63 days)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Cypress, California, United States